CLINICAL TRIAL: NCT03463369
Title: A First-In-Human, Double-Blind, Randomized, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, Reactogenicity, and Immunogenicity of JNJ-64300535, a DNA Vaccine, Administered by Electroporation-Mediated Intramuscular Injection, in Participants With Chronic Hepatitis B Who Are on Stable Nucleos(T)Ide Therapy and Virologically Suppressed
Brief Title: A First-In-Human Study to Evaluate Safety, Tolerability, Reactogenicity, and Immunogenicity of JNJ-64300535, a DNA Vaccine, Administered by Electroporation-Mediated Intramuscular Injection, in Participants With Chronic Hepatitis B Who Are on Stable Nucleos(t)Ide Therapy and Virologically Suppressed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: 64300535HPB1001; 64300535HPB1001 (Other: Janssen Sciences Ireland UC); 2017-000147-41 (EudraCT Number)
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo + Nucleos(t)ide Analogs (NA) (Experimental): Participants will receive placebo intramuscular (IM) injection on Day 1, Week 4, and Week 12, along with standard of care NA treatment.
  Interventions: Biological: Placebo; Drug: Nucleos(t)ide Analogs (NA)
- JNJ-64300535 + NA (Experimental): Participants will receive JNJ-64300535 IM injection on Day 1, Week 4, and Week 12, along with standard of care NA treatment.
  Interventions: Biological: JNJ-64300535; Drug: Nucleos(t)ide Analogs (NA)

INTERVENTIONS:
Biological: JNJ-64300535 — Participants will receive JNJ-64300535 vaccine by electroporation-mediated IM injection on Day 1, Week 4, and Week 12.
  Arms: JNJ-64300535 + NA
Biological: Placebo — Participants will receive 1 mL (0.9 percent [%] sodium chloride [NaCl]) of placebo solution matching to JNJ-64300535 electroporation-mediated IM injection on Day 1, Week 4, and Week 12.
  Arms: Placebo + Nucleos(t)ide Analogs (NA)
Drug: Nucleos(t)ide Analogs (NA) — Participants will receive NA as a standard of care treatment.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and reactogenicity of escalating doses of JNJ-64300535 delivered via electroporation-mediated intramuscular injection in nucleos(t)ide analogs (NA)-treated chronic hepatitis B (CHB) participants.

ELIGIBILITY:
Inclusion Criteria:

* Has chronic hepatitis B virus envelope antigen (HBeAg) negative hepatitis B virus (HBV) infection documented by a positive hepatitis B virus surface antigen (HBsAg) test and/or detectable HBV deoxyribonucleic acid (DNA) at least 6 months prior to the screening visit
* Is on a stable treatment with one of the approved oral nucleos(t)ide analogs (NA) polymerase inhibitors tenofovir alafenamide, tenofovir disoproxil fumarate, or entecavir for greater than or equal to (>=)12 months prior to screening. A history of switching between the above treatments is acceptable as long as it was not triggered by virologic failure
* Must demonstrate HBV DNA levels less than (<)60 international unit/milliliter (IU/mL) on 2 occasions separated by greater than (>)6 months (of which one can be the screening assessment).
* Has HBsAg levels at screening between 100 IU/mL and 10,000 IU/mL
* Has normal alanine aminotransferase (ALT) levels for at least 6 months prior to baseline with no documented measurement exceeding 1.25 times upper limit of normal [ULN]). Minimal requirement is documentation of two ALT results within the year prior to baseline of which one can be the screening assessment.

Exclusion Criteria:

* Presence of advanced hepatic fibrosis or cirrhosis in 1 of the assessments below done less than or equal to (<=)6 month prior to baseline: a. Metavir score 3 or 4 in a liver biopsy OR b. Fibroscan result of >9 kilopascal (kPa) OR c. Acoustic Radiation Force Impulse (ARFI) result of >=1.55 meter/second (m/s)
* Clinical signs or history of liver cirrhosis or hepatic decompensation:

  1. Metavir score 4 in a historical biopsy OR
  2. ascites, esophageal varices, or hepatic encephalopathy OR
  3. documentation of one of the following laboratory abnormality within 12 months of screening:

  i. direct (conjugated) bilirubin >1.2 times upper limit of normal (ULN) OR ii. prothrombin time (PT) >1.2 times ULN OR iii. serum albumin <3.5 gram per deciliter (g/dL)
* Positive serology test at screening for any of the following:

  1. anti-hepatitis B surface (ant-HBs) antibodies
  2. HBeAg
  3. anti-human immunodeficiency virus (HIV)-1 or anti-HIV-2 antibodies
  4. anti-hepatitis A virus (HAV) immunoglobulin M (IgM) antibodies
  5. anti-hepatitis C virus (ant-HCV) antibodies
  6. anti-hepatitis D virus (anti-HDV) antibodies
* Participants with any evidence of liver disease of non-HBV etiology. This includes but is not limited to hepatitis A, C, or D virus infections (as above), drug- or alcohol-related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cirrhosis, primary sclerosing cholangitis, non-alcoholic steatohepatitis or any other non-HBV liver disease considered clinically significant by the investigator
* Has a history of persistent or recurrent hyperbilirubinemia unless explained by known Gilbert's Disease
* History of blood disorders (bleeding problems or a blood clot, thalassemia major or sickle cell anemia).
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) by Severity and Relationship to Study Treatment and Dose Level | Up to Week 16
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity of AEs will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events as follows: Mild = Grade 1, Moderate = Grade 2, Severe = Grade 3, Potentially life-threatening = Grade 4.
Number of Participants With Laboratory Abnormalities | Up to Week 16
  Number of participants with laboratory abnormalities related to hematology, serum chemistry, coagulation, liver function tests and urinalysis will be reported. Laboratory abnormalities will be graded according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events as follows: Mild = Grade 1, Moderate = Grade 2, Severe = Grade 3, Potentially life-threatening = Grade 4.
Number of Participants With Clinically Significant Changes in Vital Signs | Up to Week 16
  Number of participants with clinically significant changes in the vital signs including blood pressure, pulse/heart rate, and body temperature will be reported.
Number of Participants With Clinically Significant Changes in Physical Examination (Palpation of Lymph Nodes, Height, Body Weight, and Skin Examination) Findings | Up to Week 16
  Number of participants with clinically significant changes in physical examination parameters will be reported. Full physical examination (including palpation of lymph nodes, height, body weight, and skin examination) and symptom-directed physical examination will be performed.
Number of Participants With Acute Injection Site Reactions on Day 1 | From 0 to 2 hours post-vaccination on Day 1
  Participants will be assessed for the acute injection site reactions. Acute reactions means the reactions which occur within 0 to 2 hours post-vaccination. Acute reactions will be graded as follows: Grade 0 = Normal, Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Potentially Life Threatening.
Number of Participants With Acute Injection Site Reactions at Week 4 | From 0 to 2 hours post-vaccination at Week 4
  Participants will be assessed for the acute injection site reactions. Acute reactions means the reactions which occur within 0 to 2 hours post-vaccination. Acute reactions will be graded as follows: Grade 0 = Normal, Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Potentially Life Threatening.
Number of Participants With Acute Injection Site Reactions at Week 12 | From 0 to 2 hours post-vaccination at Week 12
  Participants will be assessed for the acute injection site reactions. Acute reactions means the reactions which occur within 0 to 2 hours post-vaccination. Acute reactions will be graded as follows: Grade 0 = Normal, Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Potentially Life Threatening.
Number of Participants With Injection Site Reactions After Vaccination on Day 1 | Up to 7 days post-vaccination on Day 1
  Participants will be assessed for the Reactogenicity. Reactogenicity means injection site reactions which occur after 7 days post- vaccination. Severity of reactions will be graded as follows: Grade 0 = Normal, Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Potentially Life Threatening.
Number of Participants With Injection Site Reactions After Vaccination on Week 4 | Up to 7 days post-vaccination on Week 4
  Participants will be assessed for the Reactogenicity. Reactogenicity means injection site reactions which occur after 7 days post-vaccination. Severity of reactions will be graded as follows: Grade 0 = Normal, Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Potentially Life Threatening.
Number of Participants With Injection Site Reactions After Vaccination on Week 12 | Up to 7 days post-vaccination on Week 12
  Participants will be assessed for the Reactogenicity. Reactogenicity means injection site reactions which occur after 7 days post- vaccination. Severity of reactions will be graded as follows: Grade 0 = Normal, Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Potentially Life Threatening.

SECONDARY OUTCOMES:
Percentage of Participants With a Positive Hepatitis B Virus (HBV) Specific T Cells Response | Day 1, Week 2, 6, 14, 24, 48, and 60
  Percentage of participants with a positive HBV-specific T cells response, assessed by interferon (IFN)-gamma ELISpot assay will be reported.
Time to Detection of HBV Specific T-Cell Responses | Day 1 up to Week 60
  Time to HBV Specific T-Cell response is defined as the time interval between Day 1 (vaccination) to the date of first evidence of positive HBV Specific T-Cell response.
Percentage of CD4+ and CD8+ T-Cell Responses | Day 1, Week 2, 6, 14, 24, 48, and 60
  The activation of CD4+ and CD8+ T-cell subsets and their cytokine expression patterns (expressing at least 1 interleukin [IL]-2, tumor necrosis factor-alpha [TNF-α] or IFN-γ specific to any antigen) will be determined by Intracellular Cytokine Staining (ICS).
Hepatitis B Antigen-Specific Cellular Immune Response | Day 1, Week 2, 6, 14, 24, 48, and 60
  Magnitude of Hepatitis B antigen-specific cellular immune responses will be assessed by ICS.
Number of TriGrid Delivery System (TDS)-Intramuscular (IM) v2.0 Device Fault Conditions by Type | Day 1, Week 4 and 12
  Number of TDS-IM v2.0 device fault conditions by type will be observed. User reported fault conditions will be documented to enable assessment of the device reliability. Device functions to be assessed include electrode/needle deployment, study treatment administration, and electroporation application.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (14):
- Belgium (3):
  - ZiekenhuisNetwerk Antwerpen (ZNA) - Stuivenberg, Antwerp
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc, Brussels
  - Universite Libre de Bruxelles (ULB) - Hopital Erasme, Brussels
- Germany (6):
  - Ruprecht-Karls-U Mannheim, Mannheim, Baden-Wurttemberg
  - MH Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Essen, UK Essen, North Rhine-Westphalia
  - IFI Hamburg, Hamburg
  - UK Leipzig, Leipzig
  - Universität Regensburg, Regensburg
- United Kingdom (5):
  - Queen Elizabeth - Birmingham, Birmingham
  - Royal Free - London, London
  - King's College - London, London
  - Bart's Health - Blizard Inst. London, London
  - Pennine Acute Hospitals - Manchester, Manchester

REFERENCES:
- [Derived] Verheijden S, Conceicao-Neto N, Bourgeois S, Vandamme C, Troyer E, Kanoulas E, Maeyer D, Crabbe M, Makariadou E, Slaets L, Fevery B, Remoortere PV, Biermer M, Kennedy PTF, De Creus A. Safety, immunogenicity, and baseline immune correlates of vaccine JNJ-0535 in participants with or without CHB. NPJ Vaccines. 2026 Feb 5. doi: 10.1038/s41541-025-01364-x. Online ahead of print. PMID 41644953